CLINICAL TRIAL: NCT01314404
Title: KAP/WTP and HPV Prevalence Studies in Preparation for a Phase IV Trial of the Gardasil HPV Vaccine in a Developing World Setting (Bamako, Mali)
Brief Title: KAP/WTP and HPV Prevalence Studies in a Developing World Setting (Bamako, Mali)
Acronym: HPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Global Alliance to Immunize Against AIDS Vaccine Foundation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Anne De Groot Scientific Director, Global Alliance to Immunize Against AIDS Vaccine Foundation
Other Study IDs: HPV Study; 38433 (Other: Merck)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Human Papillomavirus
Keywords: Human papillomavirus; Prevalence; Knowledge Attitude and Practice; Willingness to Participate; Vaccine; HPV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two cervical scrapes and 2 blood samples will be collected from each of the 160 selected patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- KAP/WTP study population: The participants will range in age from 12 to 50 and will be selected randomly. The study population will be representative of the following categories: men, women, adolescent boys, and adolescent girls.
  As our study seeks to take a broad-based view of knowledge related to cervical cancer and HPV, our study population is necessarily wide-ranging. Adolescent boys and girls will be between the ages of 12 and 18; men and women will be older than 18, with at least one child that falls within the adolescent age range.
- Prevalence study population: We plan to identify and recruit women diagnosed with cervical cancer who are being treated by a doctor from the department of gynecology of the Hospital Gabriel Touré in Bamako, Mali. These patients will have been previously identified and diagnosed by clinical exam by an obstetrician-gynecologist at Gabriel Touré, and will have been identified as surgical candidates by a doctor.
  The subject has expressed a willingness to have a biopsy or other gynecological operation and have a doctor collect tissue samples during a "standard" medical appointment, has agreed to have blood drawn, was older than 18, and has the capacity to give informed consent.

SUMMARY:
The Global Alliance to Immunize Against AIDS Vaccine Foundation (GAIA Vaccine Foundation or GAIA VF) proposes to carry out a Knowledge, Attitudes, and Practices (KAP) study in conjunction with a Willingness To Participate (WTP) evaluation to establish the prevalence of cervical dysplasia, to and perform Human Papillomavirus (HPV) subtyping studies in Bamako and in Sikoro-Mekin, a village within the perimeter of Bamako, the capital of Mali, West Africa. Working with experienced collaborators, we propose to carry out an HPV prevalence study (among women diagnosed with cervical cancer at Hôpital Touré), coupled with a study of Knowledge, Attitudes and Practices (KAP) and Willingness To Participate (WTP) in an HPV vaccine study among individuals living in Sikoro-Mekin. These studies will lay the groundwork for a phase IV study of Gardasil® at the same site, which would be an important step forward for West Africa.

DETAILED DESCRIPTION:
Hypothesis:

Human Papillomavirus (HPV) vaccination with the Gardasil vaccine has the potential to eradicate cervical cancer worldwide. However, the impact of quadrivalent Gardasil vaccination in developing world settings, where HPV subtype prevalence may differ, is unknown. Prior to conducting a Phase IV trial, HPV subtyping should be studied. Furthermore, few data are available on vaccine acceptability, health systems preparedness and vaccine cost-effectiveness and long-term impact in this region of the world.

We propose to:

(i) Evaluate, in a sample of 160 women diagnosed with cervical cancer recruited from the hospital Hôpital Touré, the prevalence of HPV subtypes associated with cervical cancer. Hôpital Touré is the referral center for cervical cancer patients from the entire city of Bamako (>1.8M inhabitants).

(ii) Train local clinical staff to implement good clinical protocols and good clinical laboratory practices for cervical cancer screening, and establish HPV sub-typing methodology at the affiliated laboratory sites [Sikoro, Bamako, Mali and the National Institute for Research on Public Health (INRSP), Bamako].

(iii) Perform a survey evaluating the Knowledge Attitude and Practice (KAP) and Willingness To Participate (WTP) with regard to HPV and HPV vaccines in the proposed trials site (300 individuals will be asked to complete surveys with trained surveyors; minimum of 100 adolescents and their 200 parents). Use focus groups and house-by-house interviews as means of collecting data. Obtain information on preferred consenting, screening and notification practices.

Methodology:

(i) We plan to identify and recruit a sample of 160 women diagnosed with cervical cancer within the department of gynecology of the Hospital Gabriel Touré in Bamako, Mali. These patients will have been previously identified and diagnosed by clinical exam by an obstetrician-gynecologist at Gabriel Touré, and will have been identified as surgical candidates by a doctor. Recruitment will be done during appointments either for a curative biopsy or for a more extensive surgical procedure. No biopsy will be done just for the sake of the study. During the study, each participant will sign a consent form and undergo an interview with a nurse. The nurse will be in charge of briefly presenting the proposed study protocol and ensuring that the patient (a) had been positively diagnosed with cervical cancer (diagnoses are established from a clinical case and/or based on the patient's history), (b) voluntarily expressed a willingness to have a biopsy or other gynecological operations and have a doctor collect tissue samples during a "standard" medical appointment (i.e. not linked to the study), (c) agreed to have blood drawn, (d) was older than 18, and (e) had the capacity to give informed consent.

In order to collect the necessary data for this study, the following procedures will be used:

* Blood draws: Blood samples will be collected in order to measure antibodies against a panel of HPV types, including HPV 16 and 18. Blood samples will be sent to the laboratory for Applied Molecular Biology (LAMB/LBMA) located in Bamako, for centrifugation and serum aliquoting. The serum samples will be stored at -20°C and will be sent to the United States every four months for serological testing in the Merck laboratories.
* Serology: The serum samples will be sent to the Merck research laboratories in the United States (Wayne Laboratories) and will be tested using the Luminex immunological assay. This assay will allow for the detection of HPV types 6, 11, 16, and 18.
* Rapid test: A rapid test will be conducted on the cells from the tissue samples. This test will allow for the detection of 14 types of HPV (16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) in two and a half hours.
* Tissue collection: Two cervical scrapes will be collected from each patient. One sample will be taken of the cells on the outer opening of the cervix and the other sample will be taken of the cells inside the cervical canal. Cervical scrapes will be stored in liquid nitrogen for maximum preservation and will be sent to the Merck laboratories to be analyzed by a laboratory technician.
* HPV Polymerase Chain Reaction (PCR): PCR assays will be conducted at the Laboratory for Applied Molecular Biology (LBMA) with adherence to strict standards of good laboratory practices. HPV sub-typing will be conducted with the cells from the cervical scrapes.

In order to protect the identity and confidentiality of each patient, a unique identification number will be used. Only the study personnel - and the patient, if requested - will have access to the study results.

(ii) We will be identifying and training the experts necessary for this study. We plan to recruit and train local medical personnel in clinical and laboratory practices. We want to develop necessary protocols for this study, put an infrastructure in place, and train medical personnel. This step is necessary not only for this study, but also for preparing for a vaccine trial (if possible). The goal is to lay the groundwork for all clinical studies to come, and to improve the conditions of vaccine research in Mali.

(iii) In order to assess KAP and WTP with regard to HPV and HPV vaccines, we plan to contact the inhabitants of Sikoro-Mekin with the help of community leaders and peer educators. Sikoro is a peri-urban neighborhood of Bamako with a population of around 40,000. The study will comprise the six sectors of the neighborhood. We want to interview around 300 people total.

Two questionnaires will be given. The participant will be given the first questionnaire, which will be followed by an information and education session. This will be followed by a second, identical questionnaire that will permit us to measure information retention and comprehension from the information session. The information sessions will be conducted either in small groups or individually in order to improve the quality of information provided, as well as the contact and communication with the person being surveyed.

Data collection and analysis:

Data will be collected and analyzed according to (i) Interview and questionnaire responses (ii) HPV subtypes and (iii) serology, Polymerase Chain Reaction (PCR), and rapid test results.

Conclusion:

Conducting this study will allow us to collect information that could help bolster the fight against the spread of HPV and cervical cancer in Mali. With the development of protocols and the training of medical personnel, we are striving to reinforce human capacity, improve research conditions, and lay the groundwork for all clinical studies to come in Mali. We hope that the collection and analysis of KAP/WTP data will be used for the goal of promoting the introduction of the Gardasil vaccine in Mali. Finally in the coming years we hope to obtain approval for the use of Gardasil and to plan for an HPV vaccine trial in Mali.

ELIGIBILITY:
Inclusion Criteria:

(i) For the KAP/WTP study:

- Adolescent boys and girls must be between the ages of 12 and 18; men and women will be older than 18, with at least one child that falls within the adolescent age range. All must be residents of one of the six sectors of Mékin-Sikoro.

(ii) For the Prevalence study:

- The major eligibility criteria are that the subject is a woman who has been positively diagnosed with cervical cancer, has voluntarily expressed a willingness to have a biopsy or other gynecological operation and have a doctor collect tissue samples during a "standard" medical appointment, has agreed to have blood drawn, was older than 18, and has the capacity to give informed consent.

Exclusion Criteria:

- For the KAP/WTP study: Unwilling or unable to provide consent. Under 12 years old.

- For the Prevalence study: Male gender Women not diagnosed with cervical cancer. Under 18 years old. Unwilling or unable to provide consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: (i) The KAP/WTP study will take place in Mékin-Sikoro, a peri-urban neighborhood of Bamako with a population of around 40,000. The study will comprise the six sectors of the district, enrolling a total of 300 participants. The participants will range in age from 12 to 50 and will be selected randomly. The study population will be representative of the following categories: men, women, adolescent boys, and adolescent girls.
  (ii) The Prevalence study subjects will be recruited among women diagnosed with cervical cancer who are attending a previously arranged appointment (i.e. not linked to the study) to have either a curative biopsy or a more extensive surgical procedure with the department of gynecology at Hôpital Gabriel Touré.
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV subtypes associated with cervical cancer | 18 months
  Blood and cervicovaginal samples will be collected, for Human Papillomavirus (HPV) serotyping (serum) and Polymerase Chain Reaction (PCR) (cervicovaginal samples).
Knowledge, Attitudes and Practices (KAP) and Willingness To Participate (WTP) in an HPV vaccine study | 18 months
  Perform a survey evaluating KAP and WTP with regard to HPV and HPV vaccines in the proposed trials site.

SECONDARY OUTCOMES:
Determine usability of Gardasil in West Africa | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne De Groot, M.D., Principal Investigator — Global Alliance to Immunize Against AIDS (GAIA) Vaccine Foundation
Locations (2):
- Mali (2):
  - Community of Sikoro, Bamako, West Africa
  - Gabriel Touré Hospital, Bamako, West Africa